CLINICAL TRIAL: NCT03239470
Title: A Phase I, Open-Label, Multicenter Trial Exploring the Safety and Tolerability of Autologous Polyclonal Regulatory T Cell Therapy in Adults With Active Pemphigus (APG01)
Brief Title: Polyclonal Regulatory T Cells (PolyTregs) for Pemphigus
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of recruitment, ongoing and new feasibility issues, and the impact of the coronavirus infectious disease 19 (COVID-19) pandemic
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Autoimmunity Centers of Excellence (Other); Rho Federal Systems Division, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DAIT APG01; APG01 (Other: Autoimmunity Centers of Excellence (ACE)); NIAID CRMS ID#: 37534 (Other: DAIT NIAID)
Record Dates: First submitted 2017-08-02; First posted 2017-08-04 (Actual); Results first posted 2021-11-22 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Pemphigus Foliaceus; Pemphigus Vulgaris
Keywords: autologous polyclonal regulatory T cell therapy; PolyTregs; open-label; Phase 1 (safety)
MeSH Terms: conditions — Pemphigus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: 1.0 x 10^8 PolyTregs (Experimental): A single intravenous infusion of 1.0 x 10^8 PolyTregs will be administered.
  Interventions: Biological: Cohort 1: 1.0 x 10^8 PolyTregs
- Cohort 2: 2.5x10^8 PolyTregs (Experimental): A single intravenous infusion of 2.5x10^8 PolyTregs will be administered.
  Interventions: Biological: Cohort 2: 2.5x10^8 PolyTregs

INTERVENTIONS:
Biological: Cohort 1: 1.0 x 10^8 PolyTregs — Each participant will receive a target cell dose of 1.0 x 10^8 polyclonal Tregs.
  Other Names: Polyclonal Regulatory T Cells; autologous PolyTregs; CD4+CD127lo/negCD25+ PolyTregs
  Arms: Cohort 1: 1.0 x 10^8 PolyTregs
Biological: Cohort 2: 2.5x10^8 PolyTregs — Each participant will receive a target cell dose of 2.5x10^8 polyclonal Tregs.
  Other Names: Polyclonal Regulatory T Cells; autologous PolyTregs; CD4+CD127lo/negCD25+ PolyTregs
  Arms: Cohort 2: 2.5x10^8 PolyTregs

SUMMARY:
T cells, a type of white blood cell called a lymphocyte, play an important role in the immune system. One subtype, the regulatory T cell (Treg) helps to regulate the immune system and may provide protection against the development of autoimmune disease. The hope is that these naturally occurring Treg cells can be utilized for the treatment of autoimmune disease and potentially replace the use of chronic immunosuppressive therapies that are associated with multiple side effects. There has been a small study showing safe administration of Tregs with decreased disease activity in patients with insulin-dependent diabetes. Tregs are being studied in lupus, cancer and organ transplantation.

This phase I trial will be conducted as an open-label, dose-escalation, multicenter trial in adult participants with active pemphigus.The purpose of this study is to test the safety and effect of Treg therapy in participants who have skin (cutaneous) involvement due to pemphigus.

DETAILED DESCRIPTION:
Up to 12 adults between the ages of 18 and 75 years of age who have been diagnosed with pemphigus and meet all other entry criteria will be enrolled to receive one infusion of their own expanded Tregs at one of the following doses:

* 1.0 x 10^8 PolyTregs or
* 2.5 x 10^8 PolyTregs.

Safety, disease activity, and mechanism of action will be assessed over a three year period, using biospecimens from blood and skin. Study therapy administration will occur during an overnight stay, followed by 2 weekly visits, then monthly visits from Week 8 to Week 12, then quarterly visits from Week 26 to Week 52, then twice a year visits until Week 156.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent;
* Diagnosis of Pemphigus Vulgaris (PV) or Pemphigus Foliaceus (PF), defined by H&E staining (e.g., Haemotoxylin and Eosin) and direct immunofluorescence staining of skin biopsy at any time prior to enrollment;
* Pemphigus treated with systemic corticosteroids within the 2 years prior to screening (historic or current), or treated with rituximab ≥ 12 months prior to screening;
* Presence of:

  * anti-Dsg3 antibodies (>20.0 U/ml) at screening visit consistent with diagnosis of pemphigus vulgaris or,
  * anti-Dsg1 antibodies (>20.0 U/ml) at screening visit consistent with diagnosis of pemphigus foliaceus.
* Active of PV or PF as defined by Pemphigus Disease Area Index (PDAI) overall activity score 3-10 at screening visit, and PDAI overall activity score 1-12 at baseline visit;
* Positive test for Epstein-Barr Virus (EBV) antibody;
* Adequate venous access to support draw of 400 ml whole blood and infusion of investigational therapy; and
* An absolute Treg count of ≥ 42 cells/μL within 6 weeks prior to whole blood collection at Week -2 (i.e., 2 weeks prior to planned PolyTreg Infusion).

Exclusion Criteria:

* Initiation of systemic corticosteroid therapy, prednisone dose > 25 mg/d (or equivalent) or change in prednisone dose within 4 weeks prior to screening;
* Addition of a new medication, or change in the dose of any background medication used to treat any aspect of pemphigus within the timeframes listed below. Specifically:

  * methotrexate, mycophenolate mofetil, mycophenolic acid, azathioprine, cyclosporine or dapsone within the 6 weeks prior to screening or in the time between screening and study drug infusion,
  * intravenous Immunoglobulin (IVIG) within 12 weeks prior to screening or in the time between screening and study drug infusion (subjects on IVIG must be on stable dose for at least 12 weeks prior to screening),
  * treatment with cyclophosphamide within 12 weeks prior to screening or in the time between screening and study drug infusion.
* Doses of background medications at screening:

  * methotrexate > 25 mg/week,
  * mycophenolate mofetil > 3000 mg/d,
  * mycophenolic acid > 1080 mg/bid,
  * azathioprine > 200 mg/d,
  * cyclosporine > 2 mg/kg/d,
  * dapsone >250 mg/d,or
  * intravenous immunoglobulin (IVIG) > 4mg/kg monthly.
* Use of rituximab within the 12 months prior to screening;
* Change in dosing frequency, concentration, or applied surface area of topical steroids and/or topical calcineurin inhibitors within 2 weeks prior to screening;
* Paraneoplastic pemphigus;
* Pemphigus erythematosus;
* Pemphigus vegetans;
* Immunoglobulin A (IgA) pemphigus;
* Drug-induced pemphigus;
* Blood donation within 10 weeks prior to baseline visit (Day 0);
* Hemoglobin < 10 g/dL;
* White blood cell (WBC) count < 3,000/ mm^3 (equivalent to < 3 x10^9/L);
* Lymphocyte count < 800/mm^3 (equivalent to < 0.8 x10^9/L);
* Absolute neutrophil count < 1,500/mm^3 (equivalent to < 1.5 x10^9/L);
* Platelets < 100,000/mm^3 (equivalent to < 100 x 10^9/L);
* Liver function test [aspartate aminotransferase (AST)], alanine aminotransferase (ALT), or alkaline phosphatase (ALK)] results that are ≥ 2 times the upper limit of normal (ULN);
* Direct bilirubin > ULN;
* End stage renal disease [estimated glomerular filtration rate (eGFR) < 20 ml/min/1.73m^2 using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation];
* At or within three months of screening:

  * a positive QuantiFERON(R)-TB Gold test or positive purified protein derivative tuberculin skin test (PPD) [>5mm induration, regardless of Bacille Calmette Guerin (BCG) vaccine administration] unless completion of treatment has been documented for active Tuberculosis (TB),
  * an indeterminate QuantiFERON (R)-TB Gold test unless followed by a subsequent negative PPD or negative QuantiFERON(R)-TB Gold test as well as a consultation with and clearance by local infectious disease (ID) department.
* Recent or ongoing active bacterial, viral, fungal, or opportunistic infections requiring systemic anti-infective therapy;
* Evidence of current or prior infection with human immunodeficiency virus (HIV), hepatitis B [as assessed by HBsAg and anti-hepatitis B core antigen (HBc) Ab] or hepatitis C [as assessed by anti-Hepatitis C Virus (anti-HCV) Ab];
* Detectable circulating EBV or Cytomegalovirus (CMV) genomes or active infection;
* Chronic infection that is currently being treated with suppressive anti-infective therapy, including but not limited to tuberculosis, pneumocystis, CMV, herpes zoster, and atypical mycobacteria, with the exception of historical orolabial or localized cutaneous herpes simplex infections treated with suppressive anti- viral therapy;
* Receipt of a live-attenuated vaccine within 12 months prior to screening;
* Concomitant malignancies or a history of malignancy, with the exception of completely treated basal cell carcinoma of the skin;
* Pregnancy;
* Lactating or breastfeeding;
* Unwilling or unable to use reliable method(s) of contraception:

  * For females of child-bearing potential, from four weeks prior to Day 0 through

    1 year after Treg dosing;
  * For males, from the day of Treg infusion (baseline visit) to three months after Treg infusion.
* Use of an investigational therapeutic medication, or other biologic medications except rituximab, within the past 90 days, or 5 half-lives prior to screening, whichever is greater;
* Concomitant medical condition that places the subject at risk by participating in this study, including but not limited to:

  * another severe, systemic autoimmune disease or condition (besides pemphigus) requiring systemic immunosuppressive therapy (e.g., rheumatoid arthritis, Systemic Lupus Erythematosus (SLE), systemic sclerosis, primary Sjogren's syndrome, primary vasculitis, psoriasis, multiple sclerosis, ankylosing spondylitis, and inflammatory bowel disease), or
  * severe, progressive, or poorly controlled renal, hepatic, hematological, gastrointestinal, pulmonary, cardiac, or neurological disease, or
  * history of significant infection or recurrent infection that, in the investigator's opinion, places the subject at risk by participating in this study, or
  * any other concomitant medical condition that, in the investigator's opinion, places the subject at risk by participating in this study.
* Comorbidities requiring glucocorticoid therapy, including those which have required three or more courses of systemic glucocorticoids within the previous 12 months;
* Current or history within the past year of substance abuse; or
* Inability to comply with study and follow-up procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2023-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haley Naik, MD,MHSc, Study Chair — University of California San Francisco School of Medicine: Department of Dermatology; Anna Haemel, MD, Study Chair — University of California San Francisco School of Medicine: Department of Dermatology; Michael Rosenblum, MD, Ph.D., Study Chair — University of California San Francisco School of Medicine: Department of Dermatology; Jeffrey Bluestone, Ph.D., Study Chair — UCSF School of Medicine: UCSF Diabetes Clinic; David Wofsy, M.D., Study Chair — University of California San Francisco School of Medicine: Lupus Clinic and Rheumatology Clinical Research Center
Locations (4):
- United States (4):
  - University of California San Francisco School of Medicine: Department of Dermatology, San Francisco, California
  - University of Iowa Health Care: Department of Dermatology, Iowa City, Iowa
  - Duke University Medical Center: Department of Dermatology, Durham, North Carolina
  - University of Texas Southwestern Medical Center: Department of Dermatology, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data upon completion of the study in: Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.
Time Frame: On average, within 24 months after database lock for the trial.
Access Criteria: Open access.
URL: https://www.immport.org/home

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) website — https://www.niaid.nih.gov/about/dait
- See also: Autoimmunity Centers of Excellence (ACE) website — http://www.autoimmunitycenters.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ten participants were screened at four sites in the United States, and 5 of those participants initiated blood donation. Enrollment occurred between October 2017 and May 2020. The first participant signed informed consent on October 10, 2017.
Groups:
- Cohort 1: Polyclonal Treg Infusion (PolyTregs) Low Dose: Participants donated peripheral blood to be processed in a lab that expanded regulatory T cells (Tregs). After two weeks, participants received a single infusion of ex vivo expanded autologous CD4+CD127lo/-CD25+ polyclonal Tregs (PolyTregs). Target cell dose was 1 x 10^8 PolyTregs.
- Cohort 2: Polyclonal Treg Infusion (Poly Tregs) High Dose: Participants donated peripheral blood to be processed in a lab that expanded regulatory T cells (Tregs). After two weeks, participants received a single infusion of ex vivo expanded autologous CD4+CD127lo/-CD25+ polyclonal Tregs (PolyTregs). Target cell dose was 2.5 x 10^8 PolyTregs. Study enrollment was closed prior to enrolling participants into Cohort 2.
Period: Blood Donation
Arm/Group | Cohort 1: Polyclonal Treg Infusion (PolyTregs) Low Dose | Cohort 2: Polyclonal Treg Infusion (Poly Tregs) High Dose
Started | 5 | 0
Completed | 5 | 0
Not Completed | 0 | 0
Period: Polyclonal Treg Infusion
Arm/Group | Cohort 1: Polyclonal Treg Infusion (PolyTregs) Low Dose | Cohort 2: Polyclonal Treg Infusion (Poly Tregs) High Dose
Started | 5 (Started includes all participants who completed the pre-infusion checklist at the infusion visit. Five participants completed the pre-infusion checklist. One participant was deemed ineligible for infusion due to the baseline PDAI > 12. Four participants initiated and completed the PolyTreg infusion.) | 0
Completed | 4 (Participants who did not meet eligibility, per the pre-infusion checklist, did not complete study infusion.) | 0
Not Completed | 1 | 0
Not completed — Baseline Pemphigus Disease Area Index (PDAI) >12, thus ineligible for PolyTregs infusion. | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants who donated peripheral blood to be processed in a lab that expanded regulatory T cells (Tregs) that, after two weeks, received a single infusion of ex vivo expanded autologous CD4+CD127lo/-CD25+ polyclonal Tregs (PolyTregs). Target cell dose was 1 x 10^8 PolyTregs.
Arm/Group | Cohort 1: Polyclonal Treg Infusion (PolyTregs) Low Dose
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4
Type of Pemphigus [Count of Participants; unit: Participants] — Summary of the type of diagnosed pemphigus at screening. To be eligible for the study, participants must have diagnosis of pemphigus vulgaris or pemphigus foliaceus.
  Participants
    Pemphigus Vulgaris | 3
    Pemphigus Foliaceus | 1
Age at Diagnosis of Pemphigus [Mean (Standard Deviation); unit: years] — Study participant's age in years at the time of pemphigus diagnosis.
  years | 33.5 (16.9)

OUTCOME MEASURES:

1. Primary Outcome: Number of Significant Adverse Events Through Week 52
Description: Number of significant adverse events, defined as any related National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) version 4.03 Grade 3 or higher adverse event or any related serious adverse event (SAE). Related is defined as being possibly related or related to the ex vivo expanded autologous PolyTregs, as determined by the safety review committee.
  An SAE is any untoward medical occurrence that, at any dose* results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant.
  *Polyclonal Tregs: Ex Vivo Expanded Autologous CD4+CD127lo/-CD25+ Polyclonal Regulatory T Cells.
Time Frame: Up to Week 52
Population: Participants donated peripheral blood to be processed in a lab that expanded regulatory T cells (Tregs). After two weeks, participants received a single infusion of ex vivo expanded autologous CD4+CD127lo/-CD25+ polyclonal Tregs (PolyTregs). Target cell dose was 1 x 10^8 PolyTregs.
Measure: Number; unit: Number of Events
Groups:
- Cohort 1: Polyclonal Treg Infusion (PolyTregs): Participants donated peripheral blood to be processed in a lab that expanded regulatory T cells (Tregs). After two weeks, participants received a single infusion of ex vivo expanded autologous CD4+CD127lo/-CD25+ polyclonal Tregs (PolyTregs). Target cell dose was 1 x 10^8 PolyTregs.
Arm/Group | Cohort 1: Polyclonal Treg Infusion (PolyTregs)
Number analyzed (Participants) | 4
Number of Events | 0

2. Secondary Outcome: Number of Significant Adverse Events
Description: Number of significant adverse events, defined as any related National Cancer Institute's (NCI's) Common Toxicity Criteria for Adverse Events (CTCAE) version 4.03 Grade 3 or higher adverse event or any related serious adverse event. Related is defined as being possibly related or related to the ex vivo expanded autologous PolyTregs, as determined by the safety review committee.
Time Frame: From the start of investigational product infusion through Week 156.
Population: Participants donated peripheral blood to be processed in a lab that expanded the T cells (Tregs) to a target of 1 x 10^8 PolyTregs/mL. After two weeks, the participant was infused with their own expanded Tregs.
Measure: Number; unit: Number of Events
Groups:
- Polyclonal Treg Infusion: Participants donated peripheral blood to be processed in a lab that expanded the T cells (Tregs) to a target of 1 x 10^8 PolyTregs/mL. After two weeks, the participant was infused with their own expanded Tregs.
Arm/Group | Polyclonal Treg Infusion
Number analyzed (Participants) | 4
Number of Events | 0

3. Secondary Outcome: Number of All Adverse Events
Description: An adverse event is any untoward or unfavorable medical occurrence in a human subject, including any abnormal sign, symptom, or disease, temporally associated with the subject's participation in the research, whether or not considered related to the subject's participation in the research.
Time Frame: From the start of investigational product infusion through Week 156.
Population: as for outcome 2
Measure: Number; unit: Number of Events
Arm/Group | Polyclonal Treg Infusion
Number analyzed (Participants) | 4
Number of Events | 23

4. Secondary Outcome: Number of All NCI-CTCAE Grade 3 or Higher Adverse Events
Description: Adverse events Grade 3 or higher were graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events, Version 4.0.
Time Frame: From the start of investigational product infusion through Week 52.
Population: as for outcome 2
Measure: Number; unit: Number of Events
Arm/Group | Polyclonal Treg Infusion
Number analyzed (Participants) | 4
Number of Events | 0

5. Secondary Outcome: Number of All NCI-CTCAE Grade 3 or Higher Adverse Events
Description: as for outcome 4
Time Frame: From the start of investigational product infusion through Week 156.
Population: as for outcome 2
Measure: Number; unit: Number of Events
Arm/Group | Polyclonal Treg Infusion
Number analyzed (Participants) | 4
Number of Events | 0

6. Secondary Outcome: Number of All SAEs
Description: Number of all serious adverse events, defined as adverse events that result in the following outcomes (21 CFR 312.32(a) and ICH E2A): 1. Death 2. A life-threatening event: An AE or SAR is considered "life-threatening" if, in the view of either the investigator or DAIT, NIAID, its occurrence places the subject at immediate risk of death. It does not include an AE or SAR that, had it occurred in a more severe form, might have caused death. 3. Inpatient hospitalization or prolongation of existing hospitalization 4. Persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions 5. Congenital anomaly or birth defect 6. Important medical event that may not result in death, be life threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, it may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: From the start of investigational product infusion through Week 156.
Population: as for outcome 2
Measure: Number; unit: Number of Events
Arm/Group | Polyclonal Treg Infusion
Number analyzed (Participants) | 4
Number of Events | 0

7. Secondary Outcome: Number of All Infection Related Events
Description: If the adverse event was believed to be caused by a viral, bacterial, or fungal organism, regardless of whether it was treated with antibiotics or not, then it was classified as infection related.
Time Frame: From the start of investigational product infusion through Week 156.
Population: as for outcome 2
Measure: Number; unit: Number of Events
Arm/Group | Polyclonal Treg Infusion
Number analyzed (Participants) | 4
Number of Events | 7

8. Secondary Outcome: Number of All Infusion Reactions
Description: Defined as any adverse reaction of National Cancer Institute - Common Terminology Criteria Grade 1 and higher occurring within 24 hours of infusion. An adverse reaction means any AE caused by a drug.
Time Frame: Within 24 hours of infusion
Population: as for outcome 2
Measure: Number; unit: Number of Events
Arm/Group | Polyclonal Treg Infusion
Number analyzed (Participants) | 4
Number of Events | 5

9. Secondary Outcome: Change in Pemphigus Disease Area Index (PDAI) Score From Baseline
Description: The PDAI consists of a total activity score and a total damage score. The total activity score is a sum of the activity scores for skin, scalp and mucous membrane. The total activity score can range from 0 to 250. The total damage score is a sum of damage scores for skin and scalp. The total damage score can range from 0 to 13. Higher scores represent higher disease activity.
Time Frame: Weeks 1, 2, 8, 12, 26, 39, 52, 78, 104, 130, and 156
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Polyclonal Treg Infusion
Number analyzed (Participants) | 4
score
  PDAI Total Activity Score at Week 1 | -1.58 (1.179)
  PDAI Total Activity Score at Week 2 | -1.15 (2.845)
  PDAI Total Activity Score at Week 8 | -1.50 (3.032)
  PDAI Total Activity Score at Week 12 | -0.33 (4.392)
  PDAI Total Activity Score at Week 26 | -2.87 (3.092)
  PDAI Total Activity Score at Week 39 | -1.23 (6.823)
  PDAI Total Activity Score at Week 52 | -3.28 (3.323)
  PDAI Total Activity Score at Week 78 | -5.08 (3.496)
  PDAI Total Activity Score at Week 104 | -5.75 (4.070)
  PDAI Total Activity Score at Week 130 | -3.98 (7.617)
  PDAI Total Activity Score at Week 156 | -7.23 (2.700)
  PDAI Total Damage Score at Week 1 | 0.000 (0.816)
  PDAI Total Damage Score at Week 2 | 0.25 (1.258)
  PDAI Total Damage Score at Week 8 | -1.00 (1.414)
  PDAI Total Damage Score at Week 12 | -1.00 (1.414)
  PDAI Total Damage Score at Week 26 | -0.67 (1.155)
  PDAI Total Damage Score at Week 39 | -0.75 (0.957)
  PDAI Total Damage Score at Week 52 | -0.50 (1.291)
  PDAI Total Damage Score at Week 78 | -1.25 (1.893)
  PDAI Total Damage Score at Week 104 | -1.50 (2.380)
  PDAI Total Damage Score at Week 130 | -1.25 (2.630)
  PDAI Total Damage Score at Week 156 | -1.50 (2.380)

10. Secondary Outcome: Change in Desmoglein 1 and 3 Titers by ELISA From Baseline
Description: Autoantibodies were measured by Enzyme-Linked Immunosorbent Assays (ELISA). Blood samples were taken from participants at baseline and Weeks 1, 2, 8, 12, 26, 39, 52, 78, 104, 130, and 156. If the desmoglein 1 or desmoglein 3 titer was below the limit of detection, the lower limit of detection at the central lab was imputed. The lower limit of detection for both desmoglein 1 and desmoglein 3 was 2.5 U/mL. Change was calculated as the post-baseline value minus the baseline value. A positive difference reflects an increase in the desmoglein titer value over time; a negative difference reflects a decreased desmoglein titer over time.
Time Frame: Weeks 1, 2, 8, 12, 26, 39, 52, 78, 104, 130, and 156
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Polyclonal Treg Infusion
Number analyzed (Participants) | 4
U/mL
  Desmoglein 1 at Week 1 | 1.00 (1.414)
  Desmoglein 1 at Week 2 | 1.50 (2.082)
  Desmoglein 1 at Week 8 | -0.50 (3.873)
  Desmoglein 1 at Week 12 | 3.50 (4.123)
  Desmoglein 1 at Week 26 | -7.67 (17.786)
  Desmoglein 1 at Week 39 | -8.67 (15.144)
  Desmoglein 1 at Week 52 | -17.00 (33.237)
  Desmoglein 1 at Week 78 | -20.75 (57.968)
  Desmoglein 1 at Week 104 | -33.88 (68.940)
  Desmoglein 1 at Week 130 | -28.75 (75.168)
  Desmoglein 1 at Week 156 | -28.25 (79.943)
  Desmoglein 3 at Week 1 | -1.75 (1.708)
  Desmoglein 3 at Week 2 | -0.50 (4.123)
  Desmoglein 3 at Week 8 | 3.00 (9.309)
  Desmoglein 3 at Week 12 | 1.25 (15.457)
  Desmoglein 3 at Week 26 | 13.33 (27.538)
  Desmoglein 3 at Week 39 | -33.50 (36.919)
  Desmoglein 3 at Week 52 | -30.75 (45.966)
  Desmoglein 3 at Week 78 | -33.25 (49.789)
  Desmoglein 3 at Week 104 | -38.88 (50.150)
  Desmoglein 3 at Week 130 | -34.38 (51.406)
  Desmoglein 3 at Week 156 | -42.25 (49.291)

11. Secondary Outcome: Number of Participants Experiencing a Relapse/Flare
Description: Pemphigus relapses/flares were assessed using the consensus definition of 3 or more new lesions a month that do not heal spontaneously within 1 week or by the extension of established lesions in a patient who has achieved disease control.
Time Frame: From the start of investigational product infusion through Week 156.
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Polyclonal Treg Infusion
Number analyzed (Participants) | 4
participants | 2

12. Secondary Outcome: Time to Relapse (Flare)
Description: Pemphigus relapses/flares will be assessed using the consensus definition of 3 or more new lesions a month that do not heal spontaneously within 1 week or by the extension of established lesions in a patient who has achieved disease control. Time to flare is defined as the number of days between the date of the flare and the date of the investigational product infusion. Only participants who experienced a flare are summarized.
Time Frame: From the start of investigational product infusion through Week 156.
Population: Participants who initiated the investigational product infusion and experienced a flare between investigational product infusion and Week 156.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Polyclonal Treg Infusion
Number analyzed (Participants) | 2
Days | 149.0 (181.02)

13. Secondary Outcome: Number of Participants on Prednisone Dose ≤10 mg/Day
Description: Defined as the number of participants who were taking 0 mg/day, >0 and <=10 mg/day, or >10 mg/day of prednisone at the time of the associated study visit.
Time Frame: Weeks 12, 26, 39, 52, 78, 104, 130, and 156
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Polyclonal Treg Infusion
Number analyzed (Participants) | 4
participants
  Number taking 0 mg/day at Week 12 | 2
  Number taking >0 mg/day and <= 10 mg/day at Week 12 | 2
  Number taking >10 mg/day at Week 12 | 0
  Number taking 0 mg/day at Week 26 | 2
  Number taking >0 mg/day and <= 10 mg/day at Week 26 | 2
  Number taking >10 mg/day at Week 26 | 0
  Number taking 0 mg/day at Week 39 | 2
  Number taking >0 mg/day and <= 10 mg/day at Week 39 | 2
  Number taking >10 mg/day at Week 39 | 0
  Number taking 0 mg/day at Week 52 | 2
  Number taking >0 mg/day and <= 10 mg/day at Week 52 | 2
  Number taking >10 mg/day at Week 52 | 0
  Number taking 0 mg/day at Week 78 | 2
  Number taking >0 mg/day and <= 10 mg/day at Week 78 | 2
  Number taking >10 mg/day at Week 78 | 0
  Number taking 0 mg/day at Week 104 | 2
  Number taking >0 mg/day and <= 10 mg/day at Week 104 | 2
  Number taking >10 mg/day at Week 104 | 0
  Number taking 0 mg/day at Week 130 | 2
  Number taking >0 mg/day and <= 10 mg/day at Week 130 | 2
  Number taking >10 mg/day at Week 130 | 0
  Number taking 0 mg/day at Week 156 | 2
  Number taking >0 mg/day and <= 10 mg/day at Week 156 | 2
  Number taking >10 mg/day at Week 156 | 0

ADVERSE EVENTS:
Time Frame: Adverse Event data were collected during the following time frames: • From time of signing of informed consent until start of investigational product infusion: all SAEs • From start of investigational product infusion until 24 hours post infusion: all NCI-CTCAE Grade 1 and higher AEs • From 24 hours post-infusion until Week 52: all NCI-CTCAE Grade 2 and higher AEs • From Week 52 until Week 156: all SAEs and all NCI-CTCAE Grade 3 and higher AEs
Groups:
- Polyclonal Treg Infusion: Participants donated peripheral blood to be processed in a lab that expanded the T cells (Tregs) to 1 x 10^8 PolyTregs/mL. After two weeks, the participant was infused with their own expanded Tregs.
Arm/Group | Polyclonal Treg Infusion
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Polyclonal Treg Infusion (N=4)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
COVID-19 (Infections and infestations) | 2 (3)
Eye infection (Infections and infestations) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2)
Fascial rupture (Injury, poisoning and procedural complications) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pemphigus (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Enrollment was stopped early, on May 1, 2020, due to:

* Lack of recruitment,
* Ongoing and new feasibility issues, including the recent approval of rituximab for treatment of pemphigus, and
* The impact of the coronavirus infectious disease 19 (COVID-19) pandemic.

No participants were enrolled in Cohort 2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-17): https://cdn.clinicaltrials.gov/large-docs/70/NCT03239470/Prot_SAP_000.pdf